CLINICAL TRIAL: NCT05654623
Title: A PHASE 3, RANDOMIZED, OPEN-LABEL, MULTICENTER TRIAL OF ARV-471 (PF-07850327) VS FULVESTRANT IN PARTICIPANTS WITH ESTROGEN RECEPTOR-POSITIVE, HER2-NEGATIVE ADVANCED BREAST CANCER WHOSE DISEASE PROGRESSED AFTER PRIOR ENDOCRINE BASED TREATMENT FOR ADVANCED DISEASE (VERITAC-2)
Brief Title: A Study to Learn About a New Medicine Called Vepdegestrant (ARV-471, PF-07850327) in People Who Have Advanced Metastatic Breast Cancer
Acronym: VERITAC-2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Arvinas Estrogen Receptor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C4891001; 2022-500544-38-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2022-11-16; First posted 2022-12-16 (Actual); Results first posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Advanced Breast Cancer
Keywords: ER(+)/HER2(-) Advanced Breast Cancer; Advanced cancer of the breast; Breast neoplasm; Breast tumor; Breast cancer; Fulvestrant; Estrogen receptor positive; Metastatic breast cancer; ER degrader; PROTAC; Hormone Therapy; Hormone positive breast cancer; Endocrine therapy; Recurrent breast cancer; HR+; HER2-negative; Vepdegestrant
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ARV-471 (Experimental)
  Interventions: Drug: ARV-471
- Fulvestrant (Active Comparator)
  Interventions: Drug: Fulvestrant

INTERVENTIONS:
Drug: ARV-471 — orally, once daily on a 28-day continuous dosing schedule
  Other Names: PF-07850327
  Arms: ARV-471
Drug: Fulvestrant — intramuscularly on Days 1 and 15 of Cycle 1 and then on Day 1 of each cycle starting from C2D1 (28-day cycle)
  Arms: Fulvestrant

SUMMARY:
A study to learn about a new medicine called ARV-471 (PF-07850327) in people who have advanced metastatic breast cancer.

DETAILED DESCRIPTION:
The purpose of this study is to learn about the safety and effects of the study medicine ARV-471 (PF-07850327, vepdegestrant) compared to fulvestrant (FUL) in participants with advanced breast cancer. Advanced breast cancer is difficult to cure or control with treatment. The cancer may have spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body, i.e. bones, lungs, brain, or liver. FUL is a medicine already used for treatment of breast cancer while ARV-471 is a new medicine.

This study is seeking participants with breast cancer who:

* have cancer that has come back in the place where it started or spread to nearby tissue, lymph nodes, or distant parts of the body.
* cannot be fully cured by surgery or radiation therapy. Radiation therapy is the use of high-energy radiation such as x-rays, gamma rays and other sources to kill cancer cells and shrink tumors.
* respond to hormonal or endocrine therapy (which target hormones and/or activity of hormone receptors) such as tamoxifen or aromatase inhibitors (this is called estrogen receptor positive disease)
* have received one line of CDK4/6 inhibitor therapy (for example palbociclib, ribociclib or abemaciclib) in combination with endocrine therapy (for example letrozole) for advanced cancer.
* are allowed up to one other endocrine therapy (for example exemestane) for advanced cancer.

Half of the participants will be given ARV-471 while the other half of the participants will be given FUL.

Participants who get ARV-471 will take ARV-471 by mouth with food, one time a day. During the first treatment cycle participants who will get FUL will be given FUL by shots into the muscles on Day 1 and again 2 weeks later. After the first month, FUL shots will be given on the first day of each new treatment cycle. One treatment cycle is 28 days.

Participants will receive the study medicine until their breast cancer worsens or side effects become too severe. Participants will have visits at the study clinic about every 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants with loco-regional recurrent or metastatic breast disease not amenable to surgical resection or radiation therapy
* Confirmed diagnosis of ER+/HER2- breast cancer
* Prior therapies for locoregional recurrent or metastatic disease must fulfill all the following criteria:
* One line of CDK4/6 inhibitor therapy in combination with endocrine therapy. Only one line of CDK4/6 inhibitor is allowed in any setting.
* ≤ 1 endocrine therapy in addition to CDK4/6 inhibitor with ET
* Most recent endocrine treatment duration must have been given for ≥6 months prior to disease progression. This may be the endocrine treatment component of the CDK4/6 inhibitor line of therapy.
* Radiological progression during or after the last line of therapy.
* Measurable disease evaluable per Response Evaluation Criterion in Solid Tumors (RECIST) v.1.1 or non-measurable bone-only disease
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Participants should be willing to provide blood and tumor tissue

Exclusion Criteria:

* Participants with advanced, symptomatic visceral spread, that are at risk of life-threatening complications in the short term
* Prior treatment with:
* ARV-471, fulvestrant, elacestrant, mTOR, PI3K, AKT pathway inhibitors, PARP inhibitor for any setting
* other investigational agents (including novel endocrine therapy any SERDs, SERCAs, CERANs) for any setting
* prior chemotherapy for advanced/metastatic disease
* Inadequate liver, kidney and bone marrow function
* Active brain metastases
* Participants with significant concomitant illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 624 (Actual)
Dates: Start 2023-03-03 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2028-05-15 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (311):
- United States (87):
  - California Cancer Associates for Research and Excellence, Inc. (cCARE), Encinitas, California
  - Orange Coast Memorial Medical Center, Fountain Valley, California
  - California Cancer Associates for Research and Excellence, Fresno, California
  - Providence Queen of the Valley Medical Center, Napa, California
  - California Cancer Associates for Research and Excellence, San Marcos, California
  - Olive View-UCLA Medical Center, Sylmar, California
  - Smilow Cancer Hospital Care Center at Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital at Yale-New Haven, New Haven, Connecticut
  - Yale-New Haven Hospital, New Haven, Connecticut
  - Smilow Cancer Hospital Care Center at North Haven, North Haven, Connecticut
  - Smilow Cancer Hospital Care Center at Trumbull, Trumbull, Connecticut
  - Florida Cancer Specialists, Altamonte Springs, Florida
  - Florida Cancer Specialists BON, Bonita Springs, Florida
  - Florida Cancer Specialists BCC, Bradenton, Florida
  - Florida Cancer Specialists LRS, Bradenton, Florida
  - Florida Cancer Specialists, Brandon, Florida
  - Florida Cancer Specialists NFM, Cape Coral, Florida
  - Morton Plant Hospital - BayCare Health System, Clearwater, Florida
  - Florida Cancer Specialists, Clearwater, Florida
  - Florida Cancer Specialists, Daytona Beach, Florida
  - Florida Cancer Specialists COL, Fort Myers, Florida
  - Florida Cancer Specialists GLO, Fort Myers, Florida
  - Florida Cancer Specialists, Gainesville, Florida
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - Florida Cancer Specialists, Largo, Florida
  - Florida Cancer Specialists, Lecanto, Florida
  - Florida Cancer Specialist And Research Institute, N. Venice, Florida
  - Florida Cancer Specialists NGD, Naples, Florida
  - Florida Cnacer Specialists, North Port, Florida
  - Florida Cancer Specialists, Ocala, Florida
  - Florida Cancer Specialists, Orange City, Florida
  - Florida Cancer Specialists, Orlando, Florida
  - Florida Cancer Specialists PCH, Port Charlotte, Florida
  - Florida Cancer Specialists SAC, Sarasota, Florida
  - Florida Cancer Specialists SAD, Sarasota, Florida
  - Florida Cancer Specialists, St. Petersburg, Florida
  - Florida Cancer Specialists, Stuart, Florida
  - Florida Cancer Specialists, Tampa, Florida
  - Florida Cancer Specialists, Tavares, Florida
  - Florida Cancer Specialists, The Villages, Florida
  - Florida Cancer Specialist, Trinity, Florida
  - Florida Cancer Specialists, Vero Beach, Florida
  - Florida Cancer Specialists, Wellington, Florida
  - Florida Cancer Specialists, West Palm Beach, Florida
  - Florida Cancer Specialists, Winter Park, Florida
  - Hope and Healing Cancer Services, Hinsdale, Illinois
  - Norton Cancer Institute - Downtown, Louisville, Kentucky
  - Norton Cancer Institute, Downtown, Louisville, Kentucky
  - Norton Hospital, Louisville, Kentucky
  - Norton Cancer Institute, St Matthews Campus, Louisville, Kentucky
  - Norton Women's & Children's Hospital, Louisville, Kentucky
  - Norton Brownsboro Hospital, Louisville, Kentucky
  - Norton Cancer Institute, Brownsboro Hospital Campus, Louisville, Kentucky
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Louisiana State University Health Sciences Shreveport, Shreveport, Louisiana
  - Hattiesburg Clinic Hematology/Oncology, Hattiesburg, Mississippi
  - Mercy Clinic Oncology and Hematology, Ballwin, Missouri
  - Saint Luke's Cancer Institute, Kansas City, Missouri
  - Mercy Research - David C. Pratt Cancer Center, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - MSK Basking Ridge, Basking Ridge, New Jersey
  - MSK Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering - Bergen, Montvale, New Jersey
  - Hematology Oncology Associates of CNY, Camillus, New York
  - MSK Commack, Commack, New York
  - Hematology-Oncology Associates of Central New York, PC, East Syracuse, New York
  - MSK Westchester, Harrison, New York
  - R.J. Zuckerberg Cancer Center, Lake Success, New York
  - Northern Westchester Hospital, Mount Kisco, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - MSK Evelyn H. Lauder Breast and Imaging Center, New York, New York
  - Hematology Oncology Associates of Rockland, Nyack, New York
  - Phelps Hospital, Sleepy Hollow, New York
  - MSK Nassau, Uniondale, New York
  - Cancer Centers of Southwest Oklahoma, Lawton, Oklahoma
  - Providence Cancer Institute Franz Clinic, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - University of Virginia Health System, Charlottesville, Virginia
  - UVA Breast Care Center, Charlottesville, Virginia
  - Bon Secours Memorial Regional Medical Center, Mechanicsville, Virginia
  - Bon Secours St. Francis Medical Center, Midlothian, Virginia
  - Bon Secours St. Mary's Hospital, Richmond, Virginia
  - Providence Regional Cancer System - Aberdeen, Aberdeen, Washington
  - Providence Regional Cancer System- Centralia, Centralia, Washington
  - Providence Regional Cancer System - Lacey, Lacey, Washington
  - UW Medicine Valley Medical Center, Renton, Washington
- Argentina (10):
  - Centro de Oncología e Investigación de Buenos Aires, Berazategui, Buenos Aires
  - Instituto de Oncología Angel H. Roffo, CABA, Buenos Aires
  - Stat Research S.A., Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Fundación Cenit Para La Investigación En Neurociencias, CABA, Buenos Aires F.D.
  - Fundacion Estudios Clinicos, Rosario, Santa Fe Province
  - Sanatorio de La Mujer, Rosario, Santa Fe Province
  - Centro Oncologico Korben, Buenos Aires
  - Centro de Educación Médica e Investigaciones clínicas "Dr. Norberto Quirno" (CEMIC), Buenos Aires
  - Fundación Respirar, Buenos Aires
  - Clínica Universitaria Reina Fabiola, Córdoba
- Australia (8):
  - Coffs Harbour Health Campus, Coffs Harbour, New South Wales
  - Sunshine Coast University Private Hospital, Birtinya, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - ICON Cancer Centre - Kurralta Park, Kurralta Park, South Australia
  - Icon Cancer Centre Hobart, Hobart, Tasmania
  - Cabrini Hospital -Brighton, Brighton, Victoria
  - Barwon Health, Geelong, Victoria
  - Cabrini Hospital - Malvern, Malvern, Victoria
- Austria (2):
  - Medizinische Universität Graz, Graz, Styria
  - Uniklinikum Salzburg, Salzburg
- Belgium (5):
  - Antwerp University Hospital, Edegem, Antwerpen
  - Cliniques universitaires Saint-Luc, Woluwe-Saint-Lambert, Bruxelles-capitale, Région de
  - Grand Hôpital de Charleroi, Gilly, Hainaut
  - UZ Leuven, Leuven, Vlaams-brabant
  - Clinical Chc Montlégia, Liège
- Brazil (12):
  - Hospital Santa Rita de Cassia, Vitória, Espírito Santo
  - ONCOSITE - Centro de Pesquisa Clinica em Oncologia, Ijuí, Rio Grande do Sul
  - Centro Gaucho Integrado De Oncologia, Hematologia, Ensino E Pesquisa, Porto Alegre, Rio Grande do Sul
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Hospital São Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Centro de Pesquisa Clínica - Área Administrativa, Porto Alegre, Rio Grande do Sul
  - Hospital Mae de Deus, Porto Alegre, Rio Grande do Sul
  - ANIMI - Unidade de Tratamento Oncologico, Lages, Santa Catarina
  - Faculdade de Medicina do ABC, Santo André, São Paulo
  - A. C. Camargo Cancer Center, São Paulo, São Paulo
  - IBCC - Instituto Brasileiro de Controle do Câncer, São Paulo
  - IBCC - Núcleo de Pesquisa e Ensino, São Paulo
- Bulgaria (2):
  - Complex Oncology Center - Burgas, Burgas
  - Complex Oncology Center - Plovdiv EOOD, Plovdiv
- Canada (8):
  - Cross Cancer Institute, Edmonton, Alberta
  - BC Cancer Surrey, Surrey, British Columbia
  - The Moncton Hospital, Moncton, New Brunswick
  - Waterloo Regional Health Network, Kitchener, Ontario
  - Sunnybrook Research Institute, Toronto, Ontario
  - Unity Health Toronto, St. Michael's Hospital, Toronto, Ontario
  - Centre de Services Ambulatoires de St-Jerome, Saint-Jérôme, Quebec
  - Unité de Recherche Clinique du CISSS des Laurentides, Saint-Jérôme, Quebec
- China (32):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - Beijing Hospital, Beijing, Beijing Municipality
  - Cancer Hospital Chinese Academy of Medical Science, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou Fujian, Fujian
  - The First People's Hospital of Foshan, Foshan, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Guangxi Medical University Affiliated Tumor Hospital, Nanning, Guangxi
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The First Affiliated Hospital of Henan University of Science &Technology, Luoyang, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Wuhan Union Hospital Cancer Center, Wuhan, Hubei
  - Jinyinhu Branch of Tongji Medical College Affiliated Union Hospital, Huazhong University of Science, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Nanchang People's Hospital, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - The 2nd Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Shandong Cancer Hospital, Jinan, Shandong
  - Ruijin Hospital Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - Yunnan Province Cancer Hospital, Kunming, Yunnan
  - Sir Run Run Shaw Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - The Second Affiliated hospital of Zhejiang University school of medicine, Hangzhou, Zhejiang
  - Henan Cancer Hospital, Zhengzhou
- Czechia (3):
  - Fakultní nemocnice Brno Bohunice, Brno, Brno-město
  - Fakultni Thomayerova nemocnice, Prague, Praha 4
  - Fakultni nemocnice Kralovske Vinohrady, Prague
- Finland (3):
  - Tampereen yliopistollinen sairaala, Tampere, Pirkanmaa
  - Vaasan Keskussairaala, Vaasa, Pohjanmaa
  - Satakunnan Keskussairaala, Pori
- France (8):
  - Centre Georges François Leclerc, Dijon, Côte-d'or
  - Centre de Cancérologie du Grand Montpellier, Montpellier, Languedoc-roussillon
  - Institut de Cancérologie de l'Ouest, Saint-Herblain, Loire-atlantique
  - Institut de Cancérologie de l'Ouest, Angers, Maine-et-loire
  - Centre Jean Perrin - Centre Régional de Lutte contre le Cancer d'Auvergne, Clermont-Ferrand, Puy-de-dôme
  - Sainte Catherine Institut du Cancer Avignon Provence, Avignon, Vaucluse
  - Centre Hospitalier Universitaire de Poitiers, Poitiers, Vienne
  - Henri Mondor Hospital, Créteil, Île-de-France Region
- Onkologische Schwerpunktpraxis Kurfuerstendamm, Berlin, Germany
- Greece (5):
  - University Hospital of Patras, Pátrai, Achaḯa
  - Alexandra General Hospital of Athens, Athens, Attikí
  - Attikon General University Hospital, Chaidari/Athens, Attikí
  - University General Hospital of Heraklion, Heraklion, Irakleío
  - University General Hospital of Larissa, Larissa, Thessalía
- Hungary (2):
  - Petz Aladar Egyetemi Oktato Korhaz, Győr, Győr-Moson-Sopron
  - Budapesti Uzsoki Utcai Kórház, Budapest
- India (8):
  - Artemis hospital, Gurgaon, Haryana
  - Tata Memorial Hospital, Mumbai, Maharashtra
  - HCG Manavata Cancer Centre, Nashik, Maharashtra
  - Apex Wellness Hospital, Nashik, Maharashtra
  - Bhakti Vedanta Hospital and Research Institute, Thane, Maharashtra
  - Venkateshwar Hospital, New Delhi, National Capital Territory of Delhi
  - Rajiv Gandhi Cancer Institute And Research Centre, New Delhi, National Capital Territory of Delhi
  - Institute of Post Graduate Medical Education and Research and Seth Sukhlal Karnani Memorial Hospital, Kolkata, West Bengal
- Israel (2):
  - Rabin Medical Center, Petah Tikva, Central District
  - Kaplan Medical Center, Rehovot, Central District
- Italy (11):
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale, Napoli, Campania
  - Humanitas Istituto Clinico Catanese, Misterbianco, Catania
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Policlinico di Sant'Orsola, Bologna, Emilia-Romagna
  - Azienda Ospedaliero Universitaria di Ferrara, Cona, Ferrara
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Università Cattolica del Sacro Cuore, Rome, Lazio
  - Fondazione IRCCS San Gerardo dei Tintori, Monza, Lombardy
  - Azienda Ospedaliero Universitaria delle Marche, Ancona, The Marches
  - Azienda Ospedaliero Universitaria Pisana, Pisa, Tuscany
  - Ospedale Generale Provinciale Macerata, Macerata
  - Istituto Europeo di Oncologia IRCCS, Milan
  - Istituto Oncologico Veneto IRCCS, Padua
- Japan (18):
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Chiba cancer center, Chiba, Chiba
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - National Hospital Organization Hokkaido Cancer Center, Sapporo, Hokkaido
  - Kanagawa cancer center, Yokohama, Kanagawa
  - Osaka University Hospital, Suita, Osaka
  - Saitama Prefectural Cancer Center, Ina-machi, Saitama
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - Tokyo Metropolitan Komagome Hospital, Department of Breast Surgery, Bunkyo-ku, Tokyo
  - Cancer Institute Hospital of JFCR, Koto-ku, Tokyo
  - Japanese Foundation for Cancer Research, Koto, Tokyo
  - National Center for Global Health and Medicine, Shinjuku, Tokyo
  - Center Hospital of the National Center for Global Health and Medicine, Shinjuku-ku, Tokyo
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Sagara Hospital, Kagoshima
  - Okayama University Hospital, Okayama
- Mexico (3):
  - Boca Clinical Trials Mexico S.C., Guadajalara, Jalisco
  - Cryptex Investigación Clínica S.A. de C.V., Cuauhtémoc, Mexico City
  - Centro de Investigacion Clinica de Oaxaca, Oaxaca City
- Poland (5):
  - Centrum Badań Klinicznych Jagiellońskie Centrum Innowacji sp. z o.o., Krakow, Lesser Poland Voivodeship
  - SP ZOZ Szpital Uniwersytecki w Krakowie, Krakow, Lesser Poland Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy w Warszawie, Warsaw, Masovian Voivodeship
  - COPERNICUS PL, Wojewodzkie Centrum Onkologii, Gdansk, Pomeranian Voivodeship
  - Centrum Terapii Wspolczesnej J. M. Jasnorzewska Spolka Komandytowo-Akcyjna, Lodz, Łódź Voivodeship
- Puerto Rico (4):
  - Puerto Rico Medical Research Center, Hato Rey, Puerto RICO
  - Hospital Oncológico Dr. Isaac González-Martinez, Rio Piedras
  - Pan American Center for Oncology Trials, LLC, Rio Piedras
  - FDI Clinical Research, San Juan
- Slovakia (5):
  - Onkologicky ustav sv. Alzbety, s.r.o., Bratislava
  - Narodny onkologicky ustav, Bratislava
  - Vychodoslovensky onkologicky ustav, a.s., Košice
  - Nemocnica na okraji mesta n o, Partizánske
  - Fakultna nemocnica Trnava, Trnava
- South Africa (4):
  - Iatros International, Bloemfontein, Free State
  - Charlotte Maxeke Johannesburg Academic Hospital, Johannesburg, Gauteng
  - WCR Office, Johannesburg, Gauteng
  - Wits Clinical Research, Johannesburg, Gauteng
- South Korea (12):
  - Gachon University Gil Medical Center, Namdong-gu, Incheon-gwangyeoksi [incheon]
  - National Cancer Center, Goyang-si, Kyǒnggi-do
  - Seoul National University Bundang Hospital, Seongnam, Kyǒnggi-do
  - Ajou University Hospital, Suwon, Kyǒnggi-do
  - Korea University Anam Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - Seoul National University Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul-teukbyeolsi [seoul]
  - Asan Medical Center, Seoul, Seoul-teukbyeolsi [seoul]
  - Gangnam Severance Hospital, Yonsei University Health System, Seoul, Seoul-teukbyeolsi [seoul]
  - Samsung Medical Center, Seoul, Seoul-teukbyeolsi [seoul]
  - The Catholic Univ. of Korea Seoul St. Mary's Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - Ewha Womans University Mokdong Hospital, Seoul, Seoul-teukbyeolsi [seoul]
- Spain (19):
  - CHUAC-Hospital Teresa Herrera, A Coruña, A Coruña [LA Coruña]
  - Hospital General Universitario de Elche, Elche, Alicante
  - Institut Català d'Oncologia (ICO) - Badalona, Badalona, Barcelona [barcelona]
  - Parc de Salut Mar - Hospital del Mar, Barcelona, Barcelona [barcelona]
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [barcelona]
  - Osi Bilbao-Basurto, Bilbao, Basque Country
  - Institut Català d'Oncologia - L'Hospitalet, L'Hospitalet de Llobregat, Catalunya [cataluña]
  - Hospital Universitario Donostia, Donostia / San Sebastian, Gipuzkoa
  - Hospital Universitario Arnau de Vilanova de Lleida, Lleida, Lleida [lérida]
  - Hospital Universitario 12 de Octubre, Madrid, Madrid, Comunidad de
  - Hospital Universitario Virgen de la Victoria, Málaga, Málaga
  - Salut Sant Joan de Reus-Baix Camp (Edp), Reus, Tarragona [tarragona]
  - Hospital Universitario Virgen Nieves, Granada
  - Hospital Universitario San Cecilio, Granada
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Althaia, Xarxa Assistencial Universitària de Manresa, Manresa
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital General Universitario de Valencia, Valencia
- Södersjukhuset, Stockholm, Stockholms LÄN [se-01], Sweden
- Switzerland (3):
  - Tumor Zentrum Aarau, Aarau, Canton of Aargau
  - Kantonsspital Frauenfeld - Spital Thurgau AG, Frauenfeld, Thurgau
  - Kantonsspital Münsterlingen - Spital Thurgau AG, Münsterlingen, Thurgau
- Taiwan (12):
  - Chang Gung Memorial Hospital at Kaohsiung, Kaohsiung Niao Sung Dist, Kaohsiung
  - Chi Mei Medical Center, Tainan, Tainan
  - Chi Mei Hospital - Liouying Branch, Tainan, Tainan
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center, Taipei
  - Taipei Municipal Wan Fang Hospital, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District
- Turkey (Türkiye) (12):
  - Hacettepe Universite Hastaneleri, Altindağ, Ankara
  - TC Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi, Istanbul, İ̇stanbul
  - Acibadem Altunizade Hospital, Istanbul, İ̇stanbul
  - I.E.U. Medical Point Hastanesi, Izmir, İ̇zmir
  - Adana Medical Park Seyhan Hastanesi, Adana
  - Adana Sehir Egitim ve Arastirma Hastanesi, Adana
  - Gulhane Egitim Arastirma Hastanesi, Ankara
  - Memorial Ankara Hastanesi, Ankara
  - Ankara Bilkent Şehir Hastanesi, Ankara
  - Akdeniz Universitesi Hastanesi, Antalya
  - Trakya University Medical Faculty Hospital, Edirne
  - Samsun Medical Park Hastanesi, Samsun
- United Kingdom (4):
  - St Bartholomew's Hospital, London, London, CITY of
  - Royal Blackburn Hospital, Blackburn
  - The Beatson West of Scotland Cancer Centre, Glasgow
  - The Christie Hospital NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Campone M, De Laurentiis M, Jhaveri K, Hu X, Ladoire S, Patsouris A, Zamagni C, Cui J, Cazzaniga M, Cil T, Jerzak KJ, Fuentes C, Yoshinami T, Rodriguez-Lescure A, Sezer A, Fontana A, Guarneri V, Molckovsky A, Mouret-Reynier MA, Demirci U, Zhang Y, Valota O, Lu DR, Martignoni M, Parameswaran J, Zhi X, Hamilton EP; VERITAC-2 Study Group. Vepdegestrant, a PROTAC Estrogen Receptor Degrader, in Advanced Breast Cancer. N Engl J Med. 2025 Aug 7;393(6):556-568. doi: 10.1056/NEJMoa2505725. Epub 2025 May 31. PMID 40454645
- [Derived] Hamilton EP, Ma C, De Laurentiis M, Iwata H, Hurvitz SA, Wander SA, Danso M, Lu DR, Perkins Smith J, Liu Y, Tran L, Anderson S, Campone M. VERITAC-2: a Phase III study of vepdegestrant, a PROTAC ER degrader, versus fulvestrant in ER+/HER2- advanced breast cancer. Future Oncol. 2024;20(32):2447-2455. doi: 10.1080/14796694.2024.2377530. Epub 2024 Jul 29. PMID 39072356
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4891001

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with estrogen receptor (ER) positive, human epidermal growth factor receptor 2 negative (HER2-) unresectable locoregional recurrent or metastatic breast cancer (mBC) not amenable to radiotherapy with curative intent who progressed after prior endocrine based treatment(s) for advanced disease were included in this study.
Pre-assignment Details: Results are reported at primary completion date (31 January 2025). Remaining results will be reported on completion of analysis at study completion date.
Groups:
- Vepdegestrant (ARV-471): Participants were randomized to receive vepdegestrant 200 milligrams (mg) orally, once daily on Days 1 to 28 of each 28-day cycle. Participants continued to receive assigned treatment until objective disease progression, unacceptable toxicity, death, participant refused further treatment, or one of the other reasons for treatment discontinuation per protocol was met.
- Fulvestrant: Participants were randomized to receive fulvestrant 500 mg, intramuscularly (injection) on Days 1 and 15 of Cycle 1 and then on Day 1 of each cycle starting from Cycle 2 Day 1, where 1 cycle = 28 days. Participants continued to receive assigned treatment until objective disease progression, unacceptable toxicity, death, participant refused further treatment, or one of the other reasons for treatment discontinuation per protocol was met.
Period: Treatment
Arm/Group | Vepdegestrant (ARV-471) | Fulvestrant
Started | 313 | 311
Treated | 312 | 307
Completed | 0 | 0
Not Completed | 313 | 311
Not completed — Randomized but not treated | 1 | 4
Not completed — Adverse Event | 7 | 2
Not completed — Death | 2 | 0
Not completed — Physician Decision | 2 | 3
Not completed — Progressive disease | 189 | 209
Not completed — Protocol Violation | 2 | 0
Not completed — Withdrawal by Subject | 9 | 7
Not completed — Global deterioration of health status | 5 | 9
Not completed — Other | 0 | 1
Not completed — Ongoing | 96 | 76
Period: Follow-up
Arm/Group | Vepdegestrant (ARV-471) | Fulvestrant
Started | 205 (Participants who discontinued treatment could enter the follow-up.) | 224 (Participants who discontinued treatment could enter the follow-up.)
Completed | 0 | 0
Not Completed | 205 | 224
Not completed — Death | 43 | 35
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Ongoing | 161 | 186

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vepdegestrant (ARV-471) | Fulvestrant | Total
Number analyzed (Participants) | 313 | 311 | 624
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.3 (12.09) | 60.3 (11.52) | 60.3 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 311 | 310 | 621
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 36 | 65
  Not Hispanic or Latino | 241 | 240 | 481
  Unknown or Not Reported | 43 | 35 | 78
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 4 | 5
  Asian | 122 | 129 | 251
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 6 | 11
  White | 148 | 143 | 291
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 37 | 29 | 66

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) by Blinded Independent Central Review (BICR) Assessment Per Response Evaluation Criteria in Solid Tumors (RECIST) Version (v) 1.1- All Randomized Participants
Description: PFS assessed by BICR was defined as the time from the date of randomization to the date of the first documentation of objective progression of disease (PD) per RECIST v1.1, or death due to any cause, whichever occurred first. PD as per RECIST v1.1 was defined as at least a 20% increase in the sum of diameters of target measurable lesions above nadir (smallest sum observed considering baseline and all assessments prior to the timepoint under evaluation), with a minimum absolute increase of 5 millimeters (mm) relative to nadir or unequivocal progression of existing non-target lesions or the presence of new lesions. PFS was censored on the date of last adequate disease assessment for those who did not have a PFS event, discontinued the study treatment due to withdrawal of consent prior to an event, started a new anticancer therapy prior to an event, had an event after a gap of 2 or more missing disease assessments, or lost to follow-up. Kaplan-Meier method was used.
Time Frame: From date of randomization to date of first documentation of objective PD or death (any cause) or censoring date, whichever occurred first (up to 18.56 months and 19.38 months of treatment exposure for vepdegestrant and fulvestrant arms respectively)
Population: Full analysis set (FAS) included all enrolled participants who were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Vepdegestrant: Participants were randomized to receive vepdegestrant 200 mg orally, once daily on Days 1 to 28 of each 28-day cycle. Participants continued to receive assigned treatment until objective disease progression, unacceptable toxicity, death, participant refused further treatment, or one of the other reasons for treatment discontinuation per protocol was met.
Arm/Group | Vepdegestrant | Fulvestrant
Number analyzed (Participants) | 313 | 311
Months | 3.7 [3.6 to 5.3] | 3.6 [2.2 to 3.8]
Statistical Analysis 1: Comparison: Vepdegestrant vs Fulvestrant; Test type: Superiority; p = 0.0358, Log Rank; 1-sided P-value based on log-rank test; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.676 to 1.016] — HR was calculated based on Cox's Proportional Hazard model

2. Primary Outcome: PFS by BICR Assessment Per RECIST v1.1-Participants With ESR1 Mutation
Description: PFS assessed by BICR was defined as the time from the date of randomization to the date of the first documentation of objective PD per RECIST v1.1, or death due to any cause, whichever occurred first. PD as per RECIST v1.1 was defined as at least a 20% increase in the sum of diameters of target measurable lesions above nadir (smallest sum observed considering baseline and all assessments prior to the timepoint under evaluation), with a minimum absolute increase of 5 mm relative to nadir or unequivocal progression of existing non-target lesions or the presence of new lesions. PFS was censored on the date of last adequate disease assessment for those who did not have a PFS event, discontinued the study treatment due to withdrawal of consent prior to an event, started a new anticancer therapy prior to an event, had an event after a gap of 2 or more missing disease assessments, or lost to follow-up. Kaplan-Meier method was used.
Time Frame: as for outcome 1
Population: FAS included all enrolled participants who were randomized. Here, "Overall Number of Participants Analyzed" signifies participants with known ESR1 mutation-positive breast cancer.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Vepdegestrant | Fulvestrant
Number analyzed (Participants) | 136 | 134
Months | 5.0 [3.7 to 7.4] | 2.1 [1.9 to 3.5]
Statistical Analysis 1: Comparison: Vepdegestrant vs Fulvestrant; Test type: Superiority; p = 0.0001, Log Rank; 1-sided P-value based on log-rank test; Hazard Ratio (HR) = 0.57, 95% CI 2-sided [0.418 to 0.770] — HR was calculated based on Cox's Proportional Hazard model

3. Secondary Outcome: Overall Survival (OS)-All Randomized Participants
Description: OS was defined as the time from date of randomization to date of death due to any cause. In case of no death, OS time would be censored on the date participant was last known to be alive.
Time Frame: From date of randomization to the date of death due to any cause or censoring date
Reporting Status: Not Posted, anticipated posting 2029-05

4. Secondary Outcome: OS-Participants With ESR1 Mutation
Description: as for outcome 3
Time Frame: From date of randomization to the date of death due to any cause or censoring date
Reporting Status: Not Posted, anticipated posting 2029-05

5. Secondary Outcome: Percentage of Participants With Objective Response (OR) by BICR Assessment- Participants With Measurable Disease at Baseline
Description: OR was defined as the best overall response of confirmed complete response (CR) or partial response (PR) by BICR assessment as per RECIST v1.1 criteria. As per RECIST v1.1, CR was defined as complete disappearance of all target lesions, with the exception of nodal disease, complete disappearance of all non-target lesions and no new lesions. All nodes decreased to normal (short axis <10 mm); all target lesions and disease sites were assessed. PR was defined as at least a 30% decrease from baseline in the sum of diameters of all target lesions, non-PD/not evaluated for the non-target lesions and no new lesions. The short diameter was used in the sum for nodal target lesions, while the longest diameter was used in the sum for non-nodal target lesions, all target lesions were assessed.
Time Frame: From randomization until PD, death or start of new anticancer therapy, whichever occurred first (up to 18.56 months and 19.38 months of treatment exposure for vepdegestrant and fulvestrant arms respectively)
Population: FAS included all enrolled participants who were randomized. Here, "Overall Number of Participants Analyzed" included the participants with measurable disease at baseline (last available assessments collected on or prior to randomization date).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Vepdegestrant | Fulvestrant
Number analyzed (Participants) | 221 | 222
Percentage of participants | 10.9 [7.4 to 15.6] | 3.6 [1.8 to 6.9]

6. Secondary Outcome: Clinical Benefit Rate (CBR) by BICR Assessment
Description: CBR: percentage of participants with clinical benefit response. Clinical benefit response: confirmed CR or PR at any time, or stable disease (SD) >=24 weeks per RECIST v1.1. CR: complete disappearance of all target lesions, of all non-target lesions and no new lesions; except for nodal disease, all nodes decreased to normal (short axis <10 mm); all disease sites, all target lesions assessed. PR: >=30% decrease from baseline in sum of diameters of all target lesions, non-PD/not evaluated for non-target lesions and no new lesions; all target lesions assessed. SD: did not qualify for CR, PR, PD. All target lesions assessed. PD per RECIST v1.1: at least 20% increased sum of diameters of target measurable lesions above nadir (smallest sum observed considering baseline and all assessments prior to timepoint under evaluation), with minimum absolute increase of 5mm relative to nadir or unequivocal progression of existing non-target lesions, or new lesions.
Time Frame: From randomization until PD, death due to any cause or start of new anticancer therapy, whichever occurred first (up to 18.56 months and 19.38 months of treatment exposure for vepdegestrant and fulvestrant arms respectively)
Population: FAS included all enrolled participants who were randomized. Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Vepdegestrant | Fulvestrant
Number analyzed (Participants) | 274 | 272
Percentage of participants | 34.3 [28.9 to 40.1] | 28.7 [23.6 to 34.3]

7. Secondary Outcome: Duration of Response (DOR) by BICR Assessment
Description: DOR was defined as time from first documentation of objective tumor response (CR or PR) to first documentation of PD, or death due to any cause, whichever occurred first. CR: complete disappearance of all target lesions, of all non-target lesions and no new lesions; except for nodal disease, all nodes decreased to normal (short axis <10 mm); all disease sites, all target lesions assessed. PR: >=30% decrease from baseline in sum of diameters of all target lesions, non-PD/not evaluated for non-target lesions and no new lesions; all target lesions were assessed. The short diameter is used in the sum for nodal target lesions, while longest diameter is used in sum for non-nodal target lesions, all target lesions were assessed. DOR was analyzed in participants with an OR. PD: at least 20% increase in sum of diameters of target measurable lesions above nadir, with minimum absolute increase of 5 mm relative to nadir or unequivocal progression of existing non-target lesions, or new lesions.
Time Frame: From first documentation of objective tumor response until confirmed PD or death, whichever occurred first (up to 18.56 months and 19.38 months of treatment exposure for vepdegestrant and fulvestrant arms respectively)
Population: FAS included all enrolled participants who were randomized. Here, "Overall Number of Participants Analyzed" included the participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Vepdegestrant | Fulvestrant
Number analyzed (Participants) | 24 | 8
Months | NA [5.6 to NA] — Median and upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 7.4 [5.6 to NA] — Upper limit of 95% CI was not estimable due to insufficient number of participants with events.

8. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Treatment Emergent Serious Adverse Events (TESAEs), Treatment Related TEAEs, Grade 3 or 4 and Grade 5 TEAEs as Assessed by NCI CTCAE v5.0
Description: Adverse event (AE): any untoward medical occurrence in clinical study participant, temporally associated with use of study treatment, whether or not considered related to study treatment. AEs included both SAEs and all other (non-SAEs) AEs. SAE: any untoward medical occurrence, at any dose met one or more of following criteria: death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect or other important medical events. TEAEs: AEs that occur on or after first dose of study treatment up to 28 days after last dose of study treatment. Relatedness to study drug were judged by investigator. As per National Cancer Institute Common Terminology Criteria for AE (NCI CTCAE) severity of AEs were graded as following, Grade 1: mild, Grade 2: moderate, Grade 3: severe, Grade 4: life-threatening; urgent treatment indicated, Grade 5: death related to AE.
Time Frame: From the first dose of study treatment up to 28 days after last dose of study treatment (up to 19.56 months and 20.38 months for vepdegestrant and fulvestrant arms respectively)
Population: Safety analysis set (SAS) included all randomized participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Vepdegestrant | Fulvestrant
Number analyzed (Participants) | 312 | 307
Participants
  TEAEs | 271 | 250
  TESAEs | 32 | 28
  Treatment related TEAEs | 177 | 124
  Grade 3 or 4 TEAEs | 65 | 52
  Grade 5 TEAEs | 8 | 2

9. Secondary Outcome: Number of Participants With Grade Shift From Baseline to Maximum Post-Baseline in Hematology Parameters Assessed by NCI CTCAE v5.0
Description: Hematological parameters including neutrophil count decreased, white blood cell decreased, anemia, platelet count decreased, hemoglobin increased and leukocytosis were assessed. Baseline was defined as the last assessment on or prior to the date of the first dose of study treatment. As per NCI CTCAE v5.0, severity was graded as, Grade 1: mild, Grade 2: moderate, Grade 3: severe and Grade 4: life-threatening; urgent treatment indicated. Grade 0: Non-missing laboratory value that fell outside the grading range for the corresponding laboratory parameter. Categories with at least 1 non-zero values showing any shift in Grade from baseline to post-baseline were reported.
Time Frame: From baseline up to 28 days after last dose of study treatment (up to 19.56 months and 20.38 months for vepdegestrant and fulvestrant arms respectively)
Population: SAS included all randomized participants who receive at least 1 dose of study treatment. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Vepdegestrant (ARV-471) | Fulvestrant
Number analyzed (Participants) | 310 | 303
Participants
  Neutrophil count decreased Grade 0 to Grade 1 | 33 | 13
  Neutrophil count decreased Grade 0 to Grade 2 | 26 | 15
  Neutrophil count decreased Grade 0 to Grade 3 | 4 | 0
  Neutrophil count decreased Grade 0 to Grade 4 | 1 | 1
  Neutrophil count decreased Grade 1 to Grade 0 | 5 | 9
  Neutrophil count decreased Grade 1 to Grade 2 | 5 | 3
  Neutrophil count decreased Grade 1 to Grade 3 | 1 | 1
  Neutrophil count decreased Grade 2 to Grade 0 | 2 | 1
  Neutrophil count decreased Grade 3 to Grade 2 | 0 | 1
  White blood cell decreased Grade 0 to Grade 1 | 68 | 31
  White blood cell decreased Grade 0 to Grade 2 | 18 | 8
  White blood cell decreased Grade 0 to Grade 3 | 1 | 1
  White blood cell decreased Grade 1 to Grade 0 | 10 | 12
  White blood cell decreased Grade 1 to Grade 2 | 10 | 2
  White blood cell decreased Grade 1 to Grade 3 | 0 | 1
  White blood cell decreased Grade 2 to Grade 0 | 2 | 3
  White blood cell decreased Grade 2 to Grade 1 | 0 | 1
  Anemia Grade 0 to Grade 1 | 38 | 33
  Anemia Grade 0 to Grade 2 | 6 | 6
  Anemia Grade 0 to Grade 3 | 1 | 1
  Anemia Grade 1 to Grade 0 | 14 | 12
  Anemia Grade 1 to Grade 2 | 17 | 11
  Anemia Grade 1 to Grade 3 | 4 | 4
  Anemia Grade 2 to Grade 0 | 1 | 1
  Anemia Grade 2 to Grade 1 | 5 | 3
  Anemia Grade 2 to Grade 3 | 2 | 5
  Platelet count decreased Grade 0 to Grade 1 | 25 | 22
  Platelet count decreased Grade 0 to Grade 2 | 2 | 3
  Platelet count decreased Grade 0 to Grade 3 | 2 | 2
  Platelet count decreased Grade 1 to Grade 0 | 3 | 1
  Platelet count decreased Grade 1 to Grade 2 | 0 | 1
  Platelet count decreased Grade 1 to Grade 3 | 1 | 0
  Hemoglobin increased Grade 0 to Grade 1 | 8 | 3
  Hemoglobin increased Grade 0 to Grade 2 | 1 | 0

10. Secondary Outcome: Number of Participants With Grade Shift From Baseline to Maximum Post-Baseline in Serum Chemistry Laboratory Abnormalities Assessed by NCI CTCAE v5.0
Description: Serum chemistry parameters including alanine aminotransferase increased, alkaline phosphatase increased, aspartate aminotransferase increased, blood bilirubin increased, cholesterol high, creatinine increased, hypercalcemia, hyperkalemia, hypermagnesemia, hypernatremia, hypertriglyceridemia, hypoalbuminemia, hypocalcemia, hypoglycemia, hypokalemia, hypomagnesemia, hyponatremia were assessed. Baseline was defined as the last assessment on or prior to the date of the first dose of study treatment. As per NCI CTCAE v5.0 severity was graded as, Grade 1: mild, Grade 2: moderate, Grade 3: severe and Grade 4: life-threatening; urgent treatment indicated. Grade 0: Non-missing laboratory value that falls outside the grading range for the corresponding laboratory parameter. Categories with at least 1 non-zero values showing any shift in Grade from baseline to post-baseline were reported.
Time Frame: as for outcome 9
Population: SAS included all randomized participants who received at least 1 dose of study treatment. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure. Here, "Number Analyzed" signifies participants evaluable for the specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Vepdegestrant (ARV-471) | Fulvestrant
Number analyzed (Participants) | 310 | 303
Participants
  Alanine aminotransferase increased Grade 0 to Grade 1 | 55 | 50
  Alanine aminotransferase increased Grade 0 to Grade 2 | 6 | 5
  Alanine aminotransferase increased Grade 0 to Grade 3 | 2 | 0
  Alanine aminotransferase increased Grade 1 to Grade 0 | 52 | 72
  Alanine aminotransferase increased Grade 1 to Grade 2 | 3 | 4
  Alanine aminotransferase increased Grade 1 to Grade 3 | 0 | 3
  Alanine aminotransferase increased Grade 2 to Grade 0 | 6 | 9
  Alanine aminotransferase increased Grade 2 to Grade 1 | 1 | 0
  Alkaline phosphatase increased Grade 0 to Grade 1: number analyzed (Participants) | 310 | 302
  Alkaline phosphatase increased Grade 0 to Grade 1 | 51 | 53
  Alkaline phosphatase increased Grade 0 to Grade 2: number analyzed (Participants) | 310 | 302
  Alkaline phosphatase increased Grade 0 to Grade 2 | 1 | 5
  Alkaline phosphatase increased Grade 1 to Grade 0: number analyzed (Participants) | 310 | 302
  Alkaline phosphatase increased Grade 1 to Grade 0 | 53 | 52
  Alkaline phosphatase increased Grade 1 to Grade 2: number analyzed (Participants) | 310 | 302
  Alkaline phosphatase increased Grade 1 to Grade 2 | 8 | 7
  Alkaline phosphatase increased Grade 2 to Grade 0: number analyzed (Participants) | 310 | 302
  Alkaline phosphatase increased Grade 2 to Grade 0 | 0 | 3
  Alkaline phosphatase increased Grade 2 to Grade 1: number analyzed (Participants) | 310 | 302
  Alkaline phosphatase increased Grade 2 to Grade 1 | 0 | 1
  Alkaline phosphatase increased Grade 2 to Grade 3: number analyzed (Participants) | 310 | 302
  Alkaline phosphatase increased Grade 2 to Grade 3 | 0 | 1
  Aspartate aminotransferase increased Grade 0 to Grade 1 | 78 | 54
  Aspartate aminotransferase increased Grade 0 to Grade 2 | 2 | 4
  Aspartate aminotransferase increased Grade 0 to Grade 3 | 0 | 1
  Aspartate aminotransferase increased Grade 1 to Grade 0 | 76 | 84
  Aspartate aminotransferase increased Grade 1 to Grade 2 | 4 | 5
  Aspartate aminotransferase increased Grade 1 to Grade 3 | 5 | 4
  Aspartate aminotransferase increased Grade 2 to Grade 0 | 6 | 2
  Aspartate aminotransferase increased Grade 2 to Grade 1 | 0 | 3
  Aspartate aminotransferase increased Grade 3 to Grade 0 | 0 | 1
  Blood bilirubin increased Grade 0 to Grade 1 | 30 | 12
  Blood bilirubin increased Grade 0 to Grade 2 | 9 | 7
  Blood bilirubin increased Grade 0 to Grade 3 | 1 | 3
  Blood bilirubin increased Grade 0 to Grade 4 | 2 | 0
  Blood bilirubin increased Grade 1 to Grade 0 | 0 | 4
  Blood bilirubin increased Grade 1 to Grade 2 | 1 | 0
  Blood bilirubin increased Grade 1 to Grade 3 | 0 | 1
  Blood bilirubin increased Grade 2 to Grade 0 | 1 | 0
  Cholesterol high Grade 0 to Grade 1: number analyzed (Participants) | 273 | 263
  Cholesterol high Grade 0 to Grade 1 | 22 | 31
  Cholesterol high Grade 1 to Grade 0: number analyzed (Participants) | 273 | 263
  Cholesterol high Grade 1 to Grade 0 | 23 | 20
  Cholesterol high Grade 1 to Grade 2: number analyzed (Participants) | 273 | 263
  Cholesterol high Grade 1 to Grade 2 | 3 | 6
  Cholesterol high Grade 1 to Grade 3: number analyzed (Participants) | 273 | 263
  Cholesterol high Grade 1 to Grade 3 | 0 | 1
  Cholesterol high Grade 2 to Grade 0: number analyzed (Participants) | 273 | 263
  Cholesterol high Grade 2 to Grade 0 | 1 | 0
  Cholesterol high Grade 2 to Grade 1: number analyzed (Participants) | 273 | 263
  Cholesterol high Grade 2 to Grade 1 | 4 | 0
  Creatinine increased Grade 0 to Grade 1 | 26 | 22
  Creatinine increased Grade 0 to Grade 2 | 8 | 9
  Creatinine increased Grade 0 to Grade 3 | 0 | 1
  Creatinine increased Grade 1 to Grade 0 | 8 | 6
  Creatinine increased Grade 1 to Grade 2 | 2 | 0
  Creatinine increased Grade 1 to Grade 3 | 0 | 1
  Creatinine increased Grade 2 to Grade 1 | 0 | 1
  Hypercalcemia Grade 0 to Grade 1: number analyzed (Participants) | 310 | 302
  Hypercalcemia Grade 0 to Grade 1 | 24 | 21
  Hypercalcemia Grade 0 to Grade 2: number analyzed (Participants) | 310 | 302
  Hypercalcemia Grade 0 to Grade 2 | 2 | 0
  Hypercalcemia Grade 0 to Grade 3: number analyzed (Participants) | 310 | 302
  Hypercalcemia Grade 0 to Grade 3 | 1 | 0
  Hypercalcemia Grade 0 to Grade 4: number analyzed (Participants) | 310 | 302
  Hypercalcemia Grade 0 to Grade 4 | 1 | 0
  Hypercalcemia Grade 1 to Grade 0: number analyzed (Participants) | 310 | 302
  Hypercalcemia Grade 1 to Grade 0 | 4 | 3
  Hypercalcemia Grade 1 to Grade 2: number analyzed (Participants) | 310 | 302
  Hypercalcemia Grade 1 to Grade 2 | 1 | 0
  Hypercalcemia Grade 1 to Grade 3: number analyzed (Participants) | 310 | 302
  Hypercalcemia Grade 1 to Grade 3 | 0 | 1
  Hypercalcemia Grade 1 to Grade 4: number analyzed (Participants) | 310 | 302
  Hypercalcemia Grade 1 to Grade 4 | 1 | 1
  Hyperkalemia Grade 0 to Grade 1 | 21 | 24
  Hyperkalemia Grade 0 to Grade 2 | 4 | 3
  Hyperkalemia Grade 1 to Grade 0 | 6 | 5
  Hyperkalemia Grade 1 to Grade 2 | 1 | 0
  Hypermagnesemia Grade 0 to Grade 1: number analyzed (Participants) | 309 | 298
  Hypermagnesemia Grade 0 to Grade 1 | 10 | 9
  Hypermagnesemia Grade 0 to Grade 3: number analyzed (Participants) | 309 | 298
  Hypermagnesemia Grade 0 to Grade 3 | 1 | 0
  Hypermagnesemia Grade 1 to Grade 0: number analyzed (Participants) | 309 | 298
  Hypermagnesemia Grade 1 to Grade 0 | 2 | 3
  Hypermagnesemia Grade 3 to Grade 1: number analyzed (Participants) | 309 | 298
  Hypermagnesemia Grade 3 to Grade 1 | 0 | 1
  Hypernatremia Grade 0 to Grade 1 | 11 | 4
  Hypernatremia Grade 0 to Grade 2 | 1 | 0
  Hypernatremia Grade 1 to Grade 0 | 1 | 1
  Hypertriglyceridemia Grade 0 to Grade 1: number analyzed (Participants) | 272 | 258
  Hypertriglyceridemia Grade 0 to Grade 1 | 41 | 36
  Hypertriglyceridemia Grade 0 to Grade 2: number analyzed (Participants) | 272 | 258
  Hypertriglyceridemia Grade 0 to Grade 2 | 2 | 2
  Hypertriglyceridemia Grade 0 to Grade 3: number analyzed (Participants) | 272 | 258
  Hypertriglyceridemia Grade 0 to Grade 3 | 1 | 0
  Hypertriglyceridemia Grade 1 to Grade 0: number analyzed (Participants) | 272 | 258
  Hypertriglyceridemia Grade 1 to Grade 0 | 19 | 11
  Hypertriglyceridemia Grade 1 to Grade 2: number analyzed (Participants) | 272 | 258
  Hypertriglyceridemia Grade 1 to Grade 2 | 9 | 5
  Hypertriglyceridemia Grade 1 to Grade 3: number analyzed (Participants) | 272 | 258
  Hypertriglyceridemia Grade 1 to Grade 3 | 2 | 0
  Hypertriglyceridemia Grade 2 to Grade 0: number analyzed (Participants) | 272 | 258
  Hypertriglyceridemia Grade 2 to Grade 0 | 0 | 1
  Hypertriglyceridemia Grade 2 to Grade 1: number analyzed (Participants) | 272 | 258
  Hypertriglyceridemia Grade 2 to Grade 1 | 3 | 1
  Hypertriglyceridemia Grade 2 to Grade 3: number analyzed (Participants) | 272 | 258
  Hypertriglyceridemia Grade 2 to Grade 3 | 0 | 1
  Hypertriglyceridemia Grade 3 to Grade 4: number analyzed (Participants) | 272 | 258
  Hypertriglyceridemia Grade 3 to Grade 4 | 0 | 1
  Hypoalbuminemia Grade 0 to Grade 1: number analyzed (Participants) | 310 | 302
  Hypoalbuminemia Grade 0 to Grade 1 | 40 | 32
  Hypoalbuminemia Grade 0 to Grade 2: number analyzed (Participants) | 310 | 302
  Hypoalbuminemia Grade 0 to Grade 2 | 5 | 8
  Hypoalbuminemia Grade 1 to Grade 0: number analyzed (Participants) | 310 | 302
  Hypoalbuminemia Grade 1 to Grade 0 | 4 | 8
  Hypoalbuminemia Grade 1 to Grade 2: number analyzed (Participants) | 310 | 302
  Hypoalbuminemia Grade 1 to Grade 2 | 1 | 3
  Hypoalbuminemia Grade 1 to Grade 3: number analyzed (Participants) | 310 | 302
  Hypoalbuminemia Grade 1 to Grade 3 | 0 | 1
  Hypoalbuminemia Grade 2 to Grade 0: number analyzed (Participants) | 310 | 302
  Hypoalbuminemia Grade 2 to Grade 0 | 1 | 0
  Hypoalbuminemia Grade 2 to Grade 1: number analyzed (Participants) | 310 | 302
  Hypoalbuminemia Grade 2 to Grade 1 | 1 | 0
  Hypoalbuminemia Grade 2 to Grade 3: number analyzed (Participants) | 310 | 302
  Hypoalbuminemia Grade 2 to Grade 3 | 0 | 1
  Hypocalcemia Grade 0 to Grade 1: number analyzed (Participants) | 310 | 302
  Hypocalcemia Grade 0 to Grade 1 | 26 | 20
  Hypocalcemia Grade 0 to Grade 2: number analyzed (Participants) | 310 | 302
  Hypocalcemia Grade 0 to Grade 2 | 1 | 3
  Hypocalcemia Grade 0 to Grade 3: number analyzed (Participants) | 310 | 302
  Hypocalcemia Grade 0 to Grade 3 | 0 | 1
  Hypocalcemia Grade 1 to Grade 0: number analyzed (Participants) | 310 | 302
  Hypocalcemia Grade 1 to Grade 0 | 5 | 5
  Hypocalcemia Grade 1 to Grade 2: number analyzed (Participants) | 310 | 302
  Hypocalcemia Grade 1 to Grade 2 | 4 | 1
  Hypocalcemia Grade 2 to Grade 1: number analyzed (Participants) | 310 | 302
  Hypocalcemia Grade 2 to Grade 1 | 1 | 0
  Hypoglycemia Grade 0 to Grade 1: number analyzed (Participants) | 299 | 288
  Hypoglycemia Grade 0 to Grade 1 | 6 | 9
  Hypoglycemia Grade 0 to Grade 2: number analyzed (Participants) | 299 | 288
  Hypoglycemia Grade 0 to Grade 2 | 1 | 0
  Hypoglycemia Grade 1 to Grade 0: number analyzed (Participants) | 299 | 288
  Hypoglycemia Grade 1 to Grade 0 | 2 | 1
  Hypokalemia Grade 0 to Grade 2 | 32 | 18
  Hypokalemia Grade 0 to Grade 3 | 4 | 0
  Hypokalemia Grade 2 to Grade 0 | 0 | 1
  Hypokalemia Grade 2 to Grade 3 | 3 | 0
  Hypokalemia Grade 3 to Grade 0 | 0 | 1
  Hypomagnesemia Grade 0 to Grade 1: number analyzed (Participants) | 309 | 298
  Hypomagnesemia Grade 0 to Grade 1 | 19 | 12
  Hypomagnesemia Grade 0 to Grade 2: number analyzed (Participants) | 309 | 298
  Hypomagnesemia Grade 0 to Grade 2 | 2 | 0
  Hypomagnesemia Grade 1 to Grade 0: number analyzed (Participants) | 309 | 298
  Hypomagnesemia Grade 1 to Grade 0 | 3 | 1
  Hypomagnesemia Grade 1 to Grade 2: number analyzed (Participants) | 309 | 298
  Hypomagnesemia Grade 1 to Grade 2 | 2 | 0
  Hypomagnesemia Grade 2 to Grade 3: number analyzed (Participants) | 309 | 298
  Hypomagnesemia Grade 2 to Grade 3 | 1 | 0
  Hyponatremia Grade 0 to Grade 1 | 34 | 32
  Hyponatremia Grade 0 to Grade 3 | 4 | 2
  Hyponatremia Grade 1 to Grade 0: number analyzed (Participants) | 309 | 303
  Hyponatremia Grade 1 to Grade 0 | 7 | 8
  Hyponatremia Grade 1 to Grade 3: number analyzed (Participants) | 309 | 303
  Hyponatremia Grade 1 to Grade 3 | 1 | 0
  Hyponatremia Grade 3 to Grade 0 | 1 | 0
  Hyponatremia Grade 3 to Grade 1 | 0 | 1

11. Secondary Outcome: Number of Participants According to Categorization of Electrocardiogram (ECG) Parameters
Description: Twelve lead ECGs were collected using an automated ECG machine that calculated heart rate and measured corrected QT (QTc interval, QT interval, PR interval and QRS complex). Criteria for heart rate was as follows, <= 50 beats/minute (min), >=100 beats/min, increase from baseline >= 20 beats/min, decrease from baseline >= 20 beats/min. Criteria for PR interval was >= 220 millisecond (msec). Criteria for QRS interval was >= 120 msec. Criteria for QT interval was as follows, <=450 msec, > 450 to <= 480 msec, >480 to <=500 msec, >500 msec, increase from baseline <= 30 msec, increase from baseline > 30 to <= 60 msec. Criteria for QTCF interval was as follows, <=450 msec, > 450 to <= 480 msec, > 480 to <= 500 msec, > 500 msec, increase from baseline <= 30 msec, increase from baseline > 30 to <= 60 msec, increase from baseline > 60 msec. Baseline was defined as the last assessment on or prior to the date of the first dose of study treatment.
Time Frame: as for outcome 9
Population: SAS included all randomized participants who received at least 1 dose of study treatment. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure. Here, "Number Analyzed" signifies participants evaluable for this outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | Vepdegestrant (ARV-471) | Fulvestrant
Number analyzed (Participants) | 309 | 301
Participants
  Heart rate <= 50 beats/min | 4 | 1
  Heart rate >= 100 beats/min | 23 | 19
  Heart rate increase from baseline >=20 beats/min: number analyzed (Participants) | 307 | 301
  Heart rate increase from baseline >=20 beats/min | 17 | 15
  Heart rate decrease from baseline >=20 beats/min: number analyzed (Participants) | 307 | 301
  Heart rate decrease from baseline >=20 beats/min | 22 | 10
  PR interval >= 220 msec: number analyzed (Participants) | 305 | 301
  PR interval >= 220 msec | 4 | 4
  QRS interval >=120 msec | 6 | 10
  QT interval <=450 msec | 232 | 278
  QT interval >450 to <=480 msec | 53 | 19
  QT interval >480 to <=500 msec | 16 | 4
  QT interval > 500 msec | 8 | 0
  QT intervals increase from baseline <= 30 msec: number analyzed (Participants) | 308 | 301
  QT intervals increase from baseline <= 30 msec | 171 | 267
  QT intervals increase from baseline > 30 to <=60 msec: number analyzed (Participants) | 308 | 301
  QT intervals increase from baseline > 30 to <=60 msec | 111 | 28
  QT intervals increase from baseline > 60 msec: number analyzed (Participants) | 308 | 301
  QT intervals increase from baseline > 60 msec | 26 | 6
  QTcF interval <=450 msec: number analyzed (Participants) | 308 | 301
  QTcF interval <=450 msec | 177 | 260
  QTcF interval >450 to <=480 msec | 116 | 38
  QTcF interval >480 to <=500 msec | 11 | 1
  QTcF interval > 500 msec | 5 | 2
  QTcF interval increase from baseline <= 30 msec: number analyzed (Participants) | 307 | 301
  QTcF interval increase from baseline <= 30 msec | 228 | 291
  QTcF interval increase from baseline > 30 to <= 60 msec: number analyzed (Participants) | 307 | 301
  QTcF interval increase from baseline > 30 to <= 60 msec | 71 | 9
  QTcF interval increase from baseline > 60 msec: number analyzed (Participants) | 307 | 301
  QTcF interval increase from baseline > 60 msec | 8 | 1

12. Secondary Outcome: Number of Participants According to Categorization of QT Interval Corrected Using Fridericia's Formula (QTcF) Results-QTc Substudy Analysis Set
Description: Criteria for QTcF interval for single beat were as follows, <= 450 msec, > 450 to <= 480 msec, > 480 to <=500 msec, > 500 msec, increase from baseline <= 30 msec, increase from baseline > 30 to <= 60 msec, increase from baseline > 60 msec. Baseline was defined as the last assessment on or prior to the date of the first dose of study treatment.
Time Frame: Baseline and from the first dose of study treatment up to the end of treatment (EOT) i.e., 28 days after last dose of study treatment (approximately up to 19.56 months)
Population: QTc substudy analysis set= subset of SAS participants in vepdegestrant (ARV-471) arm, randomized at selected sites and had ECG measurements to evaluate effect of ARV-471 on QTcF via serial triplicate ECGs (centrally read), had baseline ECG measurement (Cycle 1 Day 1 pre-dose) and at least one ECG measurement on Day 1 of Cycle 2 or Cycle 3 following >= 7 consecutive days of 200 mg ARV-471. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Vepdegestrant (ARV-471)
Number analyzed (Participants) | 88
Participants
  QTcF interval for single beat <=450 msec | 63
  QTcF interval for single beat > 450 to <= 480 msec | 24
  QTcF interval for single beat >480 to <=500 msec | 0
  QTcF interval for single beat > 500 msec | 1
  QTcF interval for single beat increase from baseline <= 30 msec | 67
  QTcF interval for single beat increase from baseline >30 to <= 60 msec | 21
  QTcF interval for single beat increase from baseline > 60 msec | 0

13. Secondary Outcome: Change From Baseline in European Organization for the Research and Treatment of Cancer and Quality of Life Questionnaire (EORTC QLQ-C30) Score
Description: The EORTC QLQ-C30 contains 30 items and is composed of 5 multi-item functional scales (physical functioning, role functioning, emotional functioning, cognitive functioning and social functioning), 3 multi-item symptom scales (fatigue, pain and nausea/vomiting), 6 single item symptom scales (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial impact), and one global quality of life scale. This questionnaire contained 30 questions organized into 5 multi-item functional scales, 3 multi-item symptom scales, 6 single item symptom scales, and one global quality of life scale. All the scales and single-item measures range in score from 0 to 100. Higher scores on the functional scales represent higher levels of functioning. Higher scores on the global health status/quality of life scale represent higher health status/quality of life. Higher scores on symptom scales/items represent a greater presence of symptoms.
Time Frame: From baseline up to 28 days after last dose of study treatment
Reporting Status: Not Posted, anticipated posting 2029-05

14. Secondary Outcome: Change From Baseline in European Organization for the Research and Treatment of Cancer and Quality of Life Questionnaire-Breast Cancer Specific (EORTC QLQ-BR23) Score
Description: The EORTC QLQ-BR23 was a 23-item breast cancer-specific companion module to the EORTC-QLQ-C30 and consisted of four functional scales (body image, sexual functioning, sexual enjoyment, future perspective) and four symptom scales (systemic side-effects, breast symptoms, arm symptoms, upset by hair loss). Each item was rated by choosing 1 of 4 possible responses that record the level of intensity (1= not at all, 2= a little, 3= quite a bit, and 4= very much) within each scale. All scores are converted to a 0 to 100 scale. For functional scales, higher scores represent a better level of functioning. For symptom-oriented scales, higher scores represented greater symptom severity.
Time Frame: From baseline up to 28 days after last dose of study treatment
Reporting Status: Not Posted, anticipated posting 2029-05

15. Secondary Outcome: Change From Baseline in EuroQol 5 Dimensions 5 Level (EQ-5D-5L) Index and Visual Analogue Scale (VAS) Scores
Description: The EQ-5D-5L was a 5-item participant-completed questionnaire designed to assess health status in terms of a single index value or utility score. There were 2 components, a Health State Profile where participants rated their level of problems (1=none, 2=slight, 3=moderate, 4=severe, 5=extreme/unable) in 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), and a visual analogue scale (VAS) in which participants rated their overall health status from 0 (worst imaginable) to 100 (best imaginable). Responses to 5 dimensions comprised health state/ single utility index value. E.g. if a participant responds "no problems" for each 5 dimensions, then health state was coded as "11111" with a predefined index value to it. Every health state (coded as combination of responses) had a unique predefined utility index value assigned to it per US value sets, Overall index scores ranged from 0 to 1, with lower scores representing a higher level of dysfunction.
Time Frame: From baseline up to 28 days after last dose of study treatment
Reporting Status: Not Posted, anticipated posting 2029-05

16. Secondary Outcome: Change From Baseline in Pain Severity and Pain Interference as Assessed by Brief Pain Inventory Short Form (BPI-SF) Score
Description: The BPI-SF consisted of items to measure participant perceptions of pain severity (item 3), assess degree of interference of pain on daily functioning, body diagrams on which participants indicate location of pain, record pain medication usage, VAS assessed degree of pain relief in last 24 hours (item 9a). Items in pain severity scale evaluated pain "at its worst", "at its least", and "on average" over previous 24 hours, as well as "pain now" (at time of assessment). Participants responded on 10- point numerical rating scale, where 0 = "no pain" and 10 = "pain as bad as you can imagine". Pain interference scale asked participants to rate how their pain interferes with "enjoyment of life", "general activity", "walking ability", "mood", "sleep", "normal work" and "relations with other people." Responses for interference scale were also based on 10-points scale, where 0 = "does not interfere" and 10 = "interferes completely". Higher scores=high levels of pain, impact attributed to pain.
Time Frame: From baseline up to 28 days after last dose of study treatment
Reporting Status: Not Posted, anticipated posting 2029-05

17. Secondary Outcome: Plasma Concentration of ARV-471 and Its Epimer ARV-473
Description: Plasma concentrations of ARV-471 and its epimer ARV-473 were reported in this outcome measure.
Time Frame: Anytime between -4 to 0 hours on Day 1 of Cycle 2, Cycle 3, Cycle 5 and Cycle 7 and anytime between 5 to 7 hours on Day 1 of Cycle 2 and Cycle 3
Population: PK concentration set included all participants who were in the Safety Analysis Set and had at least 1 concentration of either ARV-471 or ARV-473. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and "Number analyzed" signifies participants evaluable for a specified timepoint.
Measure: Median (Full Range); unit: Nanograms per milliliter
Arm/Group | Vepdegestrant (ARV-471)
Number analyzed (Participants) | 288
Nanograms per milliliter
  ARV-471: Cycle 2 Day 1 (-4 to 0 hours) | 445.5 [3.05 to 1530]
  ARV-471: Cycle 2 Day 1 (5 to 7 hours): number analyzed (Participants) | 274
  ARV-471: Cycle 2 Day 1 (5 to 7 hours) | 795.5 [50.5 to 2260]
  ARV-471: Cycle 3 Day 1 (-4 to 0 hours): number analyzed (Participants) | 224
  ARV-471: Cycle 3 Day 1 (-4 to 0 hours) | 453.5 [11.5 to 1680]
  ARV-471: Cycle 3 Day 1 (5 to 7 hours): number analyzed (Participants) | 211
  ARV-471: Cycle 3 Day 1 (5 to 7 hours) | 743.0 [151 to 2170]
  ARV-471: Cycle 5 Day 1 (-4 to 0 hours): number analyzed (Participants) | 150
  ARV-471: Cycle 5 Day 1 (-4 to 0 hours) | 440.5 [0.00 to 1370]
  ARV-471: Cycle 7 Day 1 (-4 to 0 hours): number analyzed (Participants) | 104
  ARV-471: Cycle 7 Day 1 (-4 to 0 hours) | 466.0 [18.7 to 1130]
  ARV-473: Cycle 2 Day 1 (-4 to 0 hours) | 193.5 [0.00 to 628]
  ARV-473: Cycle 2 Day 1 (5 to 7 hours): number analyzed (Participants) | 274
  ARV-473: Cycle 2 Day 1 (5 to 7 hours) | 225.5 [19.3 to 700]
  ARV-473: Cycle 3 Day 1 (-4 to 0 hours): number analyzed (Participants) | 224
  ARV-473: Cycle 3 Day 1 (-4 to 0 hours) | 193.0 [6.10 to 611]
  ARV-473: Cycle 3 Day 1 (5 to 7 hours): number analyzed (Participants) | 211
  ARV-473: Cycle 3 Day 1 (5 to 7 hours) | 214.0 [26.0 to 655]
  ARV-473: Cycle 5 Day 1 (-4 to 0 hours): number analyzed (Participants) | 150
  ARV-473: Cycle 5 Day 1 (-4 to 0 hours) | 188.0 [0.00 to 561]
  ARV-473: Cycle 7 Day 1 (-4 to 0 hours): number analyzed (Participants) | 104
  ARV-473: Cycle 7 Day 1 (-4 to 0 hours) | 186.0 [10.3 to 464]

18. Secondary Outcome: Change in Plasma Circulating Tumor DNA (ctDNA) From Baseline
Description: Quantitative change in plasma ctDNA levels from baseline to each protocol specified time point (up to EOT), as assessed using a validated assay.
Time Frame: Baseline and up to EOT
Reporting Status: Not Posted, anticipated posting 2029-05

ADVERSE EVENTS:
Time Frame: Adverse events: From the first dose of study treatment up to 28 days after last dose of study treatment (up to 19.56 months and 20.38 months for vepdegestrant and fulvestrant arms respectively); All-cause mortality: From randomization until date of death due to any cause (up to 19.56 months and 20.38 months for vepdegestrant and fulvestrant arms respectively)
Description: Same event may appear as both non-SAE and SAE but are distinct events. An event may be categorized as serious in 1 participant and non-serious in another, or a participant may have experienced both SAE and non-SAE. AEs were monitored for safety analysis set. All-cause mortality was monitored for full analysis set
Arm/Group | Vepdegestrant (ARV-471) | Fulvestrant
All-Cause Mortality (participants affected / at risk) | 45/313 | 35/311
Serious Adverse Events (participants affected / at risk) | 32/312 | 28/307
Other Adverse Events (participants affected / at risk) | 233/312 | 174/307
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vepdegestrant (ARV-471) (N=312) | Fulvestrant (N=307)
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Arrhythmia (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Ischaemic enteritis (Gastrointestinal disorders) | 1 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Malignant ascites (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 3
Death (General disorders) | 1 | 0
Disease progression (General disorders) | 4 | 1
Pyrexia (General disorders) | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Dorsal ramus syndrome (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 1
Hemiparesis (Nervous system disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vepdegestrant (ARV-471) (N=312) | Fulvestrant (N=307)
Anaemia (Blood and lymphatic system disorders) | 36 | 21
Constipation (Gastrointestinal disorders) | 31 | 10
Diarrhoea (Gastrointestinal disorders) | 20 | 16
Nausea (Gastrointestinal disorders) | 42 | 27
Vomiting (Gastrointestinal disorders) | 20 | 12
Asthenia (General disorders) | 35 | 26
Fatigue (General disorders) | 49 | 23
Injection site pain (General disorders) | 0 | 26
Alanine aminotransferase increased (Investigations) | 45 | 30
Aspartate aminotransferase increased (Investigations) | 45 | 32
Blood bilirubin increased (Investigations) | 20 | 11
Electrocardiogram QT prolonged (Investigations) | 31 | 4
Neutrophil count decreased (Investigations) | 25 | 10
Weight decreased (Investigations) | 16 | 10
White blood cell count decreased (Investigations) | 21 | 7
Decreased appetite (Metabolism and nutrition disorders) | 33 | 16
Hypokalaemia (Metabolism and nutrition disorders) | 21 | 6
Hyponatraemia (Metabolism and nutrition disorders) | 16 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 33 | 33
Back pain (Musculoskeletal and connective tissue disorders) | 33 | 20
Pain in extremity (Musculoskeletal and connective tissue disorders) | 16 | 13
Headache (Nervous system disorders) | 26 | 17
Insomnia (Psychiatric disorders) | 17 | 5
Hot flush (Vascular disorders) | 22 | 19
Hypertension (Vascular disorders) | 19 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2024-11-06): https://cdn.clinicaltrials.gov/large-docs/23/NCT05654623/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-05): https://cdn.clinicaltrials.gov/large-docs/23/NCT05654623/SAP_001.pdf